CLINICAL TRIAL: NCT03582436
Title: Prospective KTD-innov Cohort of Kidney Transplants Patients
Brief Title: Rejection Diagnosis in Kidney Transplants Patients
Acronym: KTD-innov
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: K170909J; 2018-A00090-55 (Registry Identifier: IDRCB number)
Record Dates: First submitted 2018-06-25; First posted 2018-07-11 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2022-02

CONDITIONS: Kidney Transplantation; Transplant Rejection; Graft Survival
Keywords: Kidney; Allogeneic transplantation; Cohort study; Rejection; Biomarkers; Integrative medicine
MeSH Terms: conditions — Rejection, Psychology | interventions — Kidney Transplantation; Gene Expression Profiling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood samples, urines samples, kidney biopsy samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Prospective cohort: Kidney transplantation
  Interventions: Procedure: Kidney transplantation

INTERVENTIONS:
Procedure: Kidney transplantation — For the patients with the kidney transplantation, these parameters will be analysis:
  Transcriptomics analysis Characteristics of anti HLA DSA analysis Non-HLA antibodies analysis Omics blood analysis Urine chemokines analysis
  Other Names: Transcriptomics analysis; Non-HLA antibodies analysis; Omics blood analysis; Urine chemokines analysis,; Characteristics of anti HLA DSA analysis

SUMMARY:
Main objective: To constitute a prospective multicentre French cohort of kidney transplant recipients including clinical, biological and immunological evaluation combined with non-invasive biomarkers in peripheral blood and urine, and gene expression assessment in allograft biopsy in order to increase the performance of rejection diagnosis in kidney transplant patients.

the investigators hypothesise that the addition of non-invasive biomarkers and intragraft assessment of gene expression profiles will improve the diagnosis capacity of histology in kidney transplant recipients as it reveals pathophysiological pathways that are not captured by light microscopy.

DETAILED DESCRIPTION:
Rejection currently represents the major cause of allograft failure worldwide, with immediate consequences for the patients in terms of mortality, morbidity and costs for the society. The field of transplantation lacks robust assessments for immune monitoring and diagnoses. Currently, light microscopy still represents the gold standard, which has clearly been identified as imperfect. Given those facts, success of clinical trials is impaired with space for improvement of current diagnosis standards that should eventually lead to improved outcomes for kidney transplant recipients.

This study will provide the investigators with prospective data of kidney transplant patient that will allow the improvement of rejection diagnosis and individual immune monitoring for precision medicine: improvement of rejection diagnosis, stage and assessment of response to therapy. In order to estimate for each patient a probability of rejection, The investigators will generate algorithms using traditional clinical, biological and histological data that will be enriched by tissue as well as blood and urine non-invasive immune biomarkers.

These algorithms will be encapsulated in a "user-friendly" web-based application with best in-class visualisation : the TransplanScreen will display individual information with comparative and predictive context for clinicians and patients and better interfacing and communication. It will include a comprehensive TransplanScreen report based on the algorithms and included in Electronic Medical Record databases (object-oriented). It aims to provide visual and contextual information to promote personalised decision making, addressing the demand of public health authorities for improving efficiency and quality of care.

The expected benefit for participants and society will be to reduce the financial burden of graft rejection for society.

The cohort will include n=750 kidney transplant recipients in 8 French centres : 3 Parisian ones: Necker hospital, Saint-Louis Hospital and Bichat hospital and 4 regional ones: CHU Nantes, Toulouse and Bordeaux, Montpellier and Lyon Hospitals. Bichat hospital will not be recruiting but will contribute to the research.

Vulnerable participants excluded.

Schedule for the study:

* inclusion period: 12 months
* participation period (treatment - follow-up): 12 months
* total duration of the study: 24 months

Exclusion period for participation in other studies, and justification: the participation to other minimal risks and constraints studies and observational non-interventional studies is allowed during this study. There is no exclusion period at the end of study. The participation to other interventional and observational non-interventional studies is allowed after the end of the study.

Number of enrolments expected per site and per month :

* Necker Hospital: 14 patients / month
* Saint-Louis Hospital: 8 patients / month
* CHU Nantes: 10 patients / month
* Lyon Hospitals: 9 patients / month
* CHU Toulouse: 13 patients / month
* CHU Bordeaux: 9 patients / month.
* CHU Montpelier: 8/month

ELIGIBILITY:
Inclusion Criteria:

Men or female patients, Age ≥ 18 years old at the time of transplantation. Patients receiving a kidney transplant from a living or deceased donor. Patients who signed the informed consent form and willing to comply with study procedures.

Female patients of child-bearing potential must have a negative pregnancy test (serum beta-hCG) and must be practicing an effective, reliable and medically approved contraceptive regimen

Patients with a minimum weight of 40 kg

Exclusion Criteria:

History of multi-organ transplant (interference with rejection natural history).

Unable/unwilling to comply with study procedures (including foreign language speakers who are not assisted by a native French speaker).

Vulnerable participants (minors, protected adults, pregnant women, legally detained

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: New kidney transplants patients
Sampling Method: Non-Probability Sample
Enrollment: 824 (Actual)
Dates: Start 2018-06-25 (Actual); Primary Completion 2021-03-18 (Actual); Study Completion 2021-03-18 (Actual)

PRIMARY OUTCOMES:
Concordance of invasive/non-invasive biomarkers with allograft rejection | month 12
  Concordance of invasive/non-invasive biomarkers with allograft rejection diagnosed by the gold standard (histology) in kidney transplant recipients.

SECONDARY OUTCOMES:
Association of non-invasive biomarkers with different subtypes of rejection | month 12
  Association of non-invasive biomarkers with different subtypes of rejection
Association of gene sets with different subtypes of rejection in the biopsy. | month 12
  Association of gene sets with different subtypes of rejection in the biopsy.
Reclassification capacity of gene sets and non-invasive biomarkers to define allograft rejection. | month 12
  Reclassification capacity of gene sets and non-invasive biomarkers to define allograft rejection
Variation of the non-invasive biomarker signature of allograft rejection | month 12
  ariation of the non-invasive biomarker signature of allograft rejection as a response to the standard of care in kidney transplant recipients.
Variation of the gene set signature | month 12
  Variation of the gene set signature of allograft rejection from the biopsy as a response to the standard of care in kidney transplant recipients.
Cumulative incidence of antibody-mediated rejection (ABMR) | month 12
  Cumulative incidence of antibody-mediated rejection (ABMR) that occurs between D0 and M12 (ABMR that meets Banff 2015 criteria)
Cumulative incidence of T-cell-mediated rejection (TCMR) | month 12
  Cumulative incidence of T-cell-mediated rejection (TCMR) that occurs between D0 and M12 (TCMR that meets Banff 2015 criteria)
Treatment failure rate | month 12
  Treatment failure rate defined as the occurrence of 1) biopsy proven ABMR and/or TCMR, 2) graft loss, 3) patient death
Graft and patient survival | month 12
  Graft and patient survival at M6 and M12 post-transplantation
Histological evidence of ABMR and/or TCMR on protocol biopsies | month 12
  Histological evidence of ABMR and/or TCMR on protocol biopsies without other clinical findings at M3 and M12 post-transplantation
Overall pathological changes, including chronic ABMR | month 12
  Overall pathological changes, including chronic ABMR, on protocol biopsies M3 and M12 post-transplantation
Incidence of delayed graft function | month 12
  Incidence of delayed graft function (DGF) post-transplantation
Cumulative incidence and duration of dialysis. | month 12
  Cumulative incidence and duration of dialysis between 7 days and M12 post- transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Loupy, Pr, Study Director — Institut National de la Santé Et de la Recherche Médicale, France
Locations (1):
- Hopital Saint-Louis, Paris, France

REFERENCES:
- [Derived] Goutaudier V, Aubert O, Racape M, Truchot A, Sablik M, Raynaud M, Vicaut E, Rousseau O, Elias M, Divard G, Papuchon E, Danger R, Charreau B, Bouton D, Nguyen-Khoa T, Randoux-Lebrun C, Taupin JL, Gourraud PA, Giral M, Le Quintrec M, Morelon E, Couzi L, Legendre C, Lefaucheur C, Kamar N, Brouard S, Anglicheau D, Loupy A; KTD-Innov Consortium. Detection of Kidney Allograft Rejection Using Urinary Chemokines. J Am Soc Nephrol. 2025 Jun 12;36(11):2228-40. doi: 10.1681/ASN.0000000742. Online ahead of print. PMID 40504617
- [Derived] Goutaudier V, Sablik M, Racape M, Rousseau O, Audry B, Kamar N, Raynaud M, Aubert O, Charreau B, Papuchon E, Danger R, Letertre L, Couzi L, Morelon E, Le Quintrec M, Taupin JL, Vicaut E, Legendre C, Le Mai H, Potluri V, Nguyen TV, Azoury ME, Pinheiro A, Nouadje G, Sonigo P, Anglicheau D, Tieken I, Vogelaar S, Jacquelinet C, Reese P, Gourraud PA, Brouard S, Lefaucheur C, Loupy A; KTD-Innov Consortium. Design, cohort profile and comparison of the KTD-Innov study: a prospective multidimensional biomarker validation study in kidney allograft rejection. Eur J Epidemiol. 2024 May;39(5):549-564. doi: 10.1007/s10654-024-01112-w. Epub 2024 Apr 16. PMID 38625480